CLINICAL TRIAL: NCT05129293
Title: Improving Prospective Memory Via Telehealth: A Randomized Feasibility Trial
Brief Title: Improving Prospective Memory Via Telehealth
Acronym: TPMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSH 21-63
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: prospective memory; cognitive dysfunction; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Memory Intervention (Experimental): Participants randomized to the PM intervention (active group) will meet with an interventionist twice a week for four weeks. The first four sessions will focus on visual imagery, while the last four sessions will focus on implementation intentions. Participants will be led through a manualized treatment.
  Interventions: Behavioral: Prospective Memory Intervention
- Educational (Active Comparator): The control group (Education) will meet with a research assistant for the same frequency of sessions and will receive psychoeducation on MS and cognitive functioning. The interventionists will be following a manual and accompanying PowerPoint slides.
  Interventions: Behavioral: Educational

INTERVENTIONS:
Behavioral: Prospective Memory Intervention — Cognitive remediation focusing on prospective memory
  Arms: Prospective Memory Intervention
Behavioral: Educational — Psychoeducation
  Arms: Educational

SUMMARY:
Up to 70% of persons with multiple sclerosis (PwMS) experience cognitive impairment, which can have a significant impact on several aspects of their daily lives. One cognitive domain that has been shown to impact daily functioning, but is understudied in MS, is prospective memory (PM). While there have been successful PM interventions in other clinical populations, to date there has not been a specific PM intervention for PwMS that has been tested in a clinical trial.

The study will be a double-masked randomized feasibility trial, with 18 participants randomized to a PM intervention and 18 participants randomized to an active control (psychoeducation). Participants will meet with an interventionist twice a week for four weeks. Feasibility will be assessed via 1) recruitment, enrollment, and retention; 2) adherence to the treatment; 3) treatment credibility and expectancy; and 4) treatment satisfaction. A preliminary effect size (Cohen's d) will be computed for the group difference using participants' performance on the Memory for Intentions Test, which will be given at baseline (week 1) and post-treatment (week 6). Participants will also complete a battery of neuropsychological measures as part of their baseline and post-treatment assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS
* Able to read, write, and speak in English
* Between the ages of 18 and 60
* All genders
* No history of other serious neurologic or psychiatric illness, including drug or alcohol misuse
* No relapses within the past two months
* Access to the Internet and a web camera
* Not enrolled in a cognitive rehabilitation program within the past six months
* Self-reported issues "remembering places they have to be" and "things they have to do"

Exclusion Criteria:

* No diagnosis of MS
* Unable to complete the study protocol due to language barriers
* Younger than 18 or older than 61
* No gender exclusions
* History of other serious neurologic or psychiatric illness, including drug or alcohol misuse
* Had a relapse within the past two months
* No access to the Internet and/or a web camera
* Currently enrolled or enrolled in a cognitive rehabilitation program within the past six months
* No self-reported issues with "remembering places they have to be" or "things they have to do"

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Rehabilitation Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Memory Intervention | Educational
Started | 17 | 18
Completed | 15 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Memory Intervention | Educational | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.29 (9.15) | 48.17 (9.8) | 47.74 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 12 | 16 | 28
  Race: Black | 3 | 1 | 4
  Race: Multi-racial/Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Memory for Intentions Test Total Score Percentile
Description: Performance on objective prospective memory (overall performance). The MIST Total Score is calculated by summing the raw scores from the six subscales, which is transformed into percentiles using age- and education-stratified normative data. Scores ranged from <1 9 (coded as 0 for analyses) to >99 (coded as 100 for analyses), with higher scores indicating better prospective memory performance.
Time Frame: Six weeks
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Prospective Memory Intervention | Educational
Number analyzed (Participants) | 17 | 18
Percentile
  Baseline | 32.24 (21.78) | 38.94 (24.29)
  Post-Treatment | 35.02 (22.77) | 45.40 (36.62)
Statistical Analysis 1: Comparison: Prospective Memory Intervention vs Educational; Test type: Superiority; p = 0.229, ANCOVA; Adjusted for disease duration, SymptoMScreen depression and anxiety scores, and Test of Everyday Cognition baseline performance

2. Primary Outcome: Memory for Intentions Test Time Cue Subscale Percentile
Description: Performance on objective prospective memory (time-based)
Time Frame: Six weeks
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Prospective Memory Intervention | Educational
Number analyzed (Participants) | 17 | 18
Percentile
  Baseline | 35.00 (19.75) | 51.78 (24.09)
  Post-treatment | 57.89 (30.53) | 59.52 (29.89)
Statistical Analysis 1: Comparison: Prospective Memory Intervention vs Educational; Test type: Superiority; p = 0.040, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Perceived Deficits Questionnaire-Prospective Memory Subscale
Description: Subjective prospective memory. The five items in the subscale are summed, with scores ranging between 0 and 20. Higher scores indicate more subjective prospective memory issues.
Time Frame: Six weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospective Memory Intervention | Educational
Number analyzed (Participants) | 17 | 18
score on a scale
  Baseline | 10.18 (2.70) | 8.44 (2.55)
  Post-Treatment | 8.79 (2.60) | 8.30 (2.74)
Statistical Analysis 1: Comparison: Prospective Memory Intervention vs Educational; Test type: Superiority; p = 0.266, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Prospective Memory Intervention | Educational
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT05129293/Prot_SAP_000.pdf